CLINICAL TRIAL: NCT02905201
Title: A Prospective Compliance Registry for Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC) Exposed to Abiraterone Acetate (TOGETHER)
Brief Title: A Prospective Compliance Registry for Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Acronym: TOGETHER
Status: Withdrawn | Type: Observational
Why Stopped: The protocol was cancelled due timelines be not compatible with business strategy in Colombia.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108078; 212082PCR4035 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mCRPC participants: Participants will not receive any intervention as a part of this study. Participants with Metastatic Castration Resistant Prostate Cancer (mCRPC) who have adequate response to treatment (abiraterone Acetate + prednisone) will be observed to collect data for ECOG performance status, safety assessments (as described above), the collection of PROs (BPI-short form, Pain VAS, HCU questionnaire), the assessment of disease status and parameters, and the assessment of participant compliance to treatment.

SUMMARY:
The primary purpose of this study is to determine the rate of compliance to abiraterone acetate and prednisone (AA + P) treatment in Colombian Castration-resistant metastatic prostate cancer (mCRPC) participants experiencing adequate response to treatment, in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Distant metastatic disease documented by positive bone scan or metastatic lesions on computerized tomography (CT) or magnetic resonance imaging (MRI)
* Prescribed and currently (at enrollment) being treated with abiraterone acetate and prednisone (AA + P) for the treatment of Castration-resistant metastatic prostate cancer (mCRPC) according to the local product label
* Having received a minimum 1 cycle of AA + P (4 weeks), and maximum 4 consecutive cycles of AA + P (16 weeks ) prior to study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1 or 2 at enrollment

Exclusion Criteria:

* Participants who have received and terminated abiraterone acetate treatment for prostate cancer (PCa) in the past
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device less than or equal to (<=) 30 days before the start of the study or the first data collection time point
* Presence of any condition that, in the opinion of the treating physician, prohibits the participant from participating in the study or obscures the assessment of the abiraterone acetate treatment in mCRPC
* Known brain metastases
* Pathological finding consistent with small cell carcinoma of the prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in this study will be men with mCRPC currently receiving AA + P for at least 1 cycle before study enrollment, and to a maximum of 4 cycles (4 months).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Complaint With Treatment (Compliance Rate) | Month 12/ early withdrawal
  Percentage of participants who are compliant to abiraterone acetate and prednisone (AA + P) treatment in Colombian mCRPC participants experiencing adequate response to treatment will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants With Abiteraterone Acetate and Prednisone (AA + P) Treatment Suspension of mCRPC Participants Treated With AA + P | Month 12/ early withdrawal
  Treatment suspension will be defined as the interruption of drug administration (abiraterone acetate) for two or more cycles of administration.
Percentage of Participants With Abiteraterone Acetate and Prednisone (AA + P) Treatment Abandonment of mCRPC Participants Treated With AA + P | Month 12/ early withdrawal
  Treatment abandonment will be defined as patient-driven cessation of drug administration, regardless of causality.
Utilization of Health Care Resources, as Measured by the Consumption of Health Care Resources Questionnaire | Baseline, Months 3, 6, 9, 12/ early withdrawal
  Utilization of Health Care Resources will be measured by the Consumption of Health Care Resources Questionnaire, which includes questions related to the participant's use of health care resources related to Prostate cancer PCa: 1) Insurance type, 2) Extra or unscheduled visits to the study doctor, another physician/specialist, healthcare professional (like nurse, therapist, physiotherapist), 3) Admission to a hospital, 4) Visits to a hospital emergency room, 5) Use of an ambulance service, 6) Complementary alternative therapy visits.
Change From AA + P Treatment Initiation in Patient Functionality Measured by the Eastern Cooperative Oncology Group (ECOG) Scale at Baseline, Months 3, 6, 9, and 12 | AA + P treatment initiation (atleast 4 weeks prior to baseline), Baseline, Months 3, 6, 9, and 12/ early withdrawal
  ECOG is a 5-point scale 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all self-care, 3=Capable of limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no self-care, totally confined to bed or chair, 5=Dead.
Change From AA + P Treatment Initiation in Prostate-Specific Antigen (PSA) Levels at Baseline, Months 3, 6, 9, and 12 | AA + P treatment initiation (atleast 4 weeks prior to baseline), Baseline, Months 3, 6, 9, and 12/ early withdrawal
Change From AA + P Treatment Initiation in Patient Pain Assessed by the Brief Pain Inventory (BPI) at Baseline, Months 3, 6, 9, and 12 | AA + P treatment initiation (atleast 4 weeks prior to baseline), Baseline, Months 3, 6, 9, and 12/ early withdrawal
  Pain intensity was assessed by Brief Pain Inventory Short Form (BPI-sf) on 11-point numerical rating scale ranging from 0=no pain to 10=pain as bad as you can imagine.
Change From AA + P Treatment Initiation in Patient Pain Assessed by the Pain Visual Analogue Scale (VAS) at Baseline, Months 3, 6, 9, and 12 | AA + P treatment initiation (atleast 4 weeks prior to baseline), Baseline, Months 3, 6, 9, and 12/ early withdrawal
  VAS is a 100 millimeter (mm) scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain.
Change From Baseline in Patient Functionality Measured by the Eastern Cooperative Oncology Group (ECOG) Scale at Months 3, 6, 9, and 12 | Baseline, Months 3, 6, 9, 12/ early withdrawal
  ECOG is a 5-point scale 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all self-care, 3=Capable of limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no self-care, totally confined to bed or chair, 5=Dead.
Change From Baseline in Prostate-Specific Antigen (PSA) Levels at Months 3, 6, 9, and 12 | Baseline, Months 3, 6, 9, 12/ early withdrawal
Change From Baseline in Patient Pain Assessed by the Brief Pain Inventory (BPI) at Months 3, 6, 9, and 12 | Baseline, Months 3, 6, 9, 12/ early withdrawal
  Pain intensity was assessed by Brief Pain Inventory Short Form (BPI-sf) on 11-point numerical rating scale ranging from 0=no pain to 10=pain as bad as you can imagine.
Change From Baseline in Patient Pain Assessed by the Pain Visual Analogue Scale (VAS) at Months 3, 6, 9, and 12 | Baseline, Months 3, 6, 9, 12/ early withdrawal
  VAS is a 100 millimeter (mm) scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain.
Overall Survival (OS) | Month 12
  The OS is defined as the time from the date of first dose of study drug to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC